CLINICAL TRIAL: NCT01402349
Title: Chronic Rhinosinusitis in a Danish Population: Evaluation of Causes of Disease, Progress and Treatment
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Bibi Lange, Department of otorhinolaryngology, Odense University Hospital
Other Study IDs: Rhino-2010
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Rhinosinusitis
Keywords: Chronic rhinosinusitis, SNOT 22, Quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blodsamples.
Oversight: Data Monitoring Committee: No

SUMMARY:
Introduction: Chronic Rhinosinusitis (CRS) is defined as inflammation of the nose and the paranasal sinuses. It is a very common disorder increasing in both incidence and prevalence with significant impact on quality of life and substantial health care costs. In this study we evaluate the prevalence of CRS in Denmark and there is a need for consensus about diagnosing this disease. Different questionnaires and different tests used for examination are evaluated together with the patients compliance and days lost through illness.

Methods: As part of Ga2len (Global Asthma and Allergy European Network) a questionnaire on CRS was posted to 5000 residents on Funen. From the completed and returned questionnaires self reported CRS was evaluated. Respondents were invited for clinical examination including spirometry, skin prick test, bloodsample and an ENT examination including nasal endoscopy, acoustic rhinometry, peak nasal inspiratory flow and smell test. Questionnaire on quality of life (EQ-5D) and symptom severity (SNOT-22) was completed. Medical diagnosed CRS was diagnosed according to the definition on CRS stated by EPOS (European Position Paper on Rhinosinusitis and Nasal Polyps 2007). CRS is defined as inflammation in the nose and paranasal sinus and should be characterized by two or more symptoms one of which should be either nasal blockage/obstruction/congestion or nasal discharge, +/- facial pain/pressure, +/- reduction or loss of smell. Endoscopic signs should be present and symptoms must have been present > 12 weeks. Patients diagnosed with CRS were invited for a 1 year and 2 year follow up where examination and questionnaires were repeated and treatment compliance and days lost through illness were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* residents on Funen aged 18-75 years

Exclusion Criteria:

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As part of Ga2len (Global Asthma and Allergy European Network) a questionnaire on CRS was posted to 5000 residents on Funen. From the completed and returned questionnaires self reported CRS was evaluated. Respondents were invited for clinical examination. Patients diagnosed with CRS were invited for a 1 year and 2 year follow up.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bibi Lange, MD, Principal Investigator — Department of Otorhinolaryngology, Odense University Hospital